CLINICAL TRIAL: NCT01124656
Title: A One-Year Phase 3, Open-Label Study to Evaluate the Safety and Tolerability of AD 4833-536 in Subjects With Type 2 Diabetes
Brief Title: Safety and Tolerability of Pioglitazone-Azilsartan in Subjects With Type 2 Diabetes
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Formulation issues.
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-06-TL-OPI536-005; U1111-1114-6658 (Registry Identifier: WHO)
Record Dates: First submitted 2010-05-13; First posted 2010-05-17 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: angiotensin II receptor blocker; thiazolidinediones; combination; Actos; HbA1c; Type 2 diabetes; Drug Therapy; Hypertension
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension | interventions — Pioglitazone; azilsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pioglitazone-Azilsartan QD (Experimental): (Dependent on glycosylated hemoglobin level at screening)
  Interventions: Drug: Pioglitazone-Azilsartan

INTERVENTIONS:
Drug: Pioglitazone-Azilsartan — Pioglitazone-Azilsartan (30 mg + 20 mg) or (45 mg + 20 mg), tablets, orally, once daily for up to 52 weeks.
  Other Names: Pioglitazone; Actos; Azilsartan; AD-4833; TAK-536

SUMMARY:
The purpose of this study is to determine the safety and tolerability of pioglitazone-azilsartan, once daily (QD), in patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
AD-4833-536 is a combination of AD-4833 (pioglitazone) and TAK-536 (azilsartan). Pioglitazone is an oral antidiabetic agent that acts by reducing insulin resistance and approved for treatment of adult patients with type 2 diabetes mellitus. Azilsartan is a angiotensin II receptor blocker that modulates the renin-angiotensin-aldosterone system that regulates blood pressure. In a recent clinical trial conducted in subjects with moderately poor to poor control of their type 2 diabetes mellitus, azilsartan coadministered with pioglitazone showed a reduction in hemoglobin A1C and fasting plasma glucose levels.

After a one week screening period, subjects will be stratified to receive a starting dose of pioglitazone-azilsartan (30 mg + 20 mg or 45 mg + 20 mg).

The planned open-label treatment period was 52 weeks; however due to formulation issues, the study was prematurely discontinued and efficacy data were not analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Has type 2 diabetes with glycosylated hemoglobin ≥7.0 % to ≤ 11.0% at Screening.
* Has been on a stable diabetic diet/exercise program.
* If receiving anti-glycemic therapy, he/she must be on ≤ two (2) anti-glycemic agents and be on a stable regimen for a minimum of 8 weeks prior to Screening.
* Has clinical laboratory evaluations at Screening (including clinical chemistry, hematology, and complete urinalysis) within the reference range for the testing laboratory unless the results are deemed not clinically significant for inclusion into this study by the investigator.
* A female subject of childbearing potential who is sexually active agrees to use adequate contraception from screening throughout the duration of the study.

Exclusion Criteria:

* Currently taking or is expected to take thiazolidinediones within 12 weeks of Screening.
* Hypersensitive to thiazolidinediones.
* Hypertension with diastolic blood pressure >100 mm Hg and/or systolic blood pressure >170 mm Hg at Screening and/or Visit 2 (Day 1).
* Currently taking an angiotensin II-receptor blocker (ARB) and is not willing to discontinue therapy at Visit 2 (day 1) and remain off for the duration of the study.
* Hypersensitive to angiotensin II-receptor blocker.
* Unstable angina or heart failure of any etiology with New York Heart Association functional class III or IV.
* History of myocardial infarction, cerebrovascular accident , percutaneous coronary intervention, coronary artery bypass graft or transient ischemic attack within the previous six months.
* Clinically significant cardiac conduction defects
* Body mass index >45 kg/m2 at Screening.
* Moderate to severe renal dysfunction
* Anemia
* Hematuria (>1+ blood) at Screening.
* Triglycerides >600 mg/dL at Screening.
* Hyperkalemia, defined as serum potassium level of greater than the upper limit of normal, per the central laboratory at Screening.
* Alanine aminotransferase or aspartate aminotransferase level of greater than 2.5 times the upper limit of normal, active liver disease, or jaundice at Screening.
* History of drug abuse or a history of alcohol abuse within the past 2 years.
* Previous history of cancer, other than basal cell carcinoma or stage 1 squamous cell carcinoma of the skin, that has not been in remission for at least 5 years prior to the first dose of study drug.
* Any other serious disease or condition that would compromise subject safety, might affect life expectancy, or make it difficult to successfully manage and follow the subject according to the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-09; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events. | On Occurrence (up to 52 Weeks).
  The Incidence of Treatment-Emergent Adverse Events, with an incidence > 5%.

SECONDARY OUTCOMES:
Change from Baseline for Glycosylated Hemoglobin. | Baseline and Weeks 4, 8, 12, 16, 24, 32, 40, 48 and 52.
  The change between the value of Glycosylated Hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at each week indicated including final visit, and Glycosylated Hemoglobin collected at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: VP, Clinical Science, Study Director — Takeda

REFERENCES:
- See also: ACTOS® Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ACTOSPI